CLINICAL TRIAL: NCT03247816
Title: Feraccru® Real World Effectiveness Study in Hospital Practice (FRESH): A Real World Study to Describe the Outcomes Associated With the Use of Ferric Maltol (Feraccru) for the Management of Iron Deficiency Anaemia in Patients With Inflammatory Bowel Disease in the UK.
Brief Title: Feraccru® Real World Effectiveness Study in Hospital Practice ( FRESH )
Acronym: FRESH
Status: Completed | Type: Observational
Sponsor: Shield Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ST10-01-401
Record Dates: First submitted 2017-03-12; First posted 2017-08-14 (Actual); Results first posted 2020-09-25 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Anemia, Iron Deficiency; Inflammatory Bowel Diseases
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to understand the early experiences of Feraccru® in patients with inflammatory bowel disease (IBD) and iron deficiency anaemia (IDA) in the UK, including treatment effectiveness, patterns of use and tolerability.

DETAILED DESCRIPTION:
The aim of the study is to understand the early experiences of Feraccru® in patients with inflammatory bowel disease (IBD) and iron deficiency anaemia (IDA) in the UK, including treatment effectiveness, patterns of use and tolerability. By describing the characteristics of patients treated with Feraccru® and their outcomes, this study will provide the medical community with important information to support treatment decisions for their patients. This will ultimately support improvements to patient care, including the long-term outcomes of patients with IBD and IDA

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥ 18 years at the time of initiation .
* Patient presenting with mild to moderate IDA that is secondary to either Crohn's disease (CD) or ulcerative colitis (UC) defined as Hb ≥9.5 g/dL and <13.0 g/dL in males, or Hb ≥9.5 g/dL and <12.0 g/dL in females
* Serum ferritin concentration <30 microgram/L or transferrin saturation of <20% .
* Patient receiving Feraccru® since the time of UK launch in June 2016.

Exclusion Criteria:

* Patient receiving Feraccru® as part of an interventional clinical trial.
* Patients with severely active IBD or requiring corticosteroids at the time of initiation on Feraccru®.
* Patient with an IBD flare, as determined by the clinician.
* Patient with medical records that are not available for review.
* Patient not willing or unable to consent to study participation, or patient is deceased at the start of data collection period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real World subjects with IBD (Crohn's disease or ulcerative colitis) who are also diagnosed with mild-moderate IDA.
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Southampton General Hospital, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Number of Eligible Subjects: Number of eligible subjects following the initial invitation to collect data on retrospective and prospective data.
Period: Overall Study
Arm/Group | Number of Eligible Subjects
Started | 59
Completed | 30
Not Completed | 29
Not completed — Adverse Event | 12
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 10
Not completed — Missing Feraccru stop date | 3

BASELINE CHARACTERISTICS:
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Age, Customized [Count of Participants; unit: Participants]
  18 < 25 | 8
  25 < 35 | 16
  35 < 45 | 12
  45 < 55 | 8
  55 < 65 | 5
  >65 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 21
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 59
Baseline Haemoglobin [Mean (Standard Deviation); unit: g/dl] | 11.1 (0.9)
Type of Inflammatory Bowel Disease [Count of Participants; unit: Participants]
  Crohn's Disease (CD) | 28
  Ulcerative Colitis (UC) | 28
  Unspecified | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Patients With Normalised Hb Levels at 12 Weeks After Initiation of Feraccru®.
Description: Normalised haemoglobin is defined in this study as Hb ≥12.0 g/dL for females and and (≥13.0 g/dL for males.
Time Frame: 12 weeks (permitting 10-16 weeks)
Population: Number of subjects with Hb measurement at 12 weeks (permitting 10-16 weeks) following initiation with Feraccru.
Measure: Count of Participants; unit: Participants
Groups:
- Normalised Hb at 12 Weeks: Normalisation of haemoglobin at 12 weeks (permitting 10-16 weeks) after initiation of Feraccru.
- Not Normalised Hb at 12 Weeks: Not normalised haemoglobin result at 12 weeks (permitting 10-16 weeks) after initiation of Feraccru.
Arm/Group | Normalised Hb at 12 Weeks | Not Normalised Hb at 12 Weeks
Number analyzed (Participants) | 30 | 30
Participants | 19 | 11

2. Secondary Outcome: Change in Hb Levels at Week 4
Description: Change in Haemoglobin levels from baseline to Week 4
Time Frame: Baseline to Week 4 (permitting 3 to 5 weeks)
Population: Subjects with available Hb at Week 4 (permitting 3 to 5 weeks).
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 17
g/dl | 0.8 (0.8)

3. Secondary Outcome: Change in Hb Levels at 12 Weeks
Description: Change in Haemoglobin levels from baseline to Week 12
Time Frame: Baseline to Week 12 (permitting 10-16 weeks)
Population: Subjects with available Hb at Week 12 (permitting 10-16 weeks).
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 30
g/dl | 1.4 (1.7)

4. Secondary Outcome: Time to Normalisation of Hb Levels
Description: Normalised haemoglobin is defined in this study as Hb ≥12.0 g/dL for females and ≥13.0 g/dL for males.
Time Frame: Baseline to 12 weeks (permitting 10-16 weeks)
Population: Subjects with available Hb at Week 12 (permitting 10-16 weeks)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 30
days | 49.5 (25.6)

5. Secondary Outcome: Change in Serum Ferritin Levels at Week 4
Description: Change in serum ferritin levels from baseline to week 4
Time Frame: Baseline to Week 4 (permitting 3 to 5 weeks)
Population: Subjects with available ferritin measurements at Week 4 (permitting 3 to 5 weeks).
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 7
ug/ml | 11.9 (12.5)

6. Secondary Outcome: Change in Serum Ferritin Levels at Week 12
Description: Change in serum ferritin levels from baseline to week 12
Time Frame: Baseline to Week 12 (permitting 10-16 weeks)
Population: Subjects with available ferritin measurement at Week 12 (permitting 10-16 weeks)
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 17
ug/ml | 19.1 (36.0)

7. Secondary Outcome: Percentage of Patients With Normalised Ferritin Levels at 12 Weeks
Description: Normalised serum ferritin is defined in this study as serum ferritin concentration ≥30 microgram/L and ≤300 microgram/L.
Time Frame: Baseline to Week 12 (permitting 10-16 weeks)
Population: Subjects with available ferritin measurements at Week 12 (permitting 10-16 weeks).
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 22
Participants | 9

8. Secondary Outcome: Time to Correction of Serum Ferritin Levels
Description: Normalised serum ferritin is defined in this study as serum ferritin concentration ≥30 microgram/L and ≤300 microgram/L.
Time Frame: Baseline to Week 12 (permitting 10 to 16 weeks)
Population: Subjects with available ferritin measurement at Week 12 (permitting 10 to 16 weeks).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 16
days | 68.0 (25.1)

9. Secondary Outcome: Change in Transferrin Saturation at Week 4
Description: Change in transferrin saturation (TSAT) at Week 4
Time Frame: Baseline to Week 4 (permitting 3 to 5 weeks)
Population: Due to insufficient data, this outcome could not be measured.
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Transferrin Saturation at Week 12
Description: Change in transferrin saturation (TSAT) at Week 12
Time Frame: Baseline to Week 12
Population: Due to insufficient data, this outcome could not be measured.
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Patients With Normalised Transferrin Saturation at 12 Weeks After Initiation of Feraccru®
Description: Normalised transferrin saturation is defined in this study as transferrin saturation between 20% and 50%.
Time Frame: Baseline to Week 12
Population: Due to insufficient data, this outcome could not be measured.
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 0

12. Secondary Outcome: Time to Correction of Transferrin Saturation
Description: Normalised transferrin saturation is defined in this study as transferrin saturation between 20% and 50%.
Time Frame: Baseline to Week 12
Population: Due to insufficient data, this outcome could not be measured.
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 0

13. Secondary Outcome: Time From Diagnosis of IBD to Initiation of Feraccru
Description: Time from diagnosis of Inflammatory Bowel Disease to initiation of Feraccru.
Time Frame: Baseline
Population: Subjects with available medical history on IBD prior to Feraccru.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 56
years | 9.4 (9.7)

14. Secondary Outcome: Time From Diagnosis of IDA to Initiation of Feraccru®
Description: Time from diagnosis of Iron Deficiency Anaemia to initiation of Feraccru®
Time Frame: Baseline
Population: Subjects with available medical history on IDA prior to Feraccru.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 54
days | 53.8 (110.4)

15. Secondary Outcome: Prior IV Treatment History
Description: Prior intravenous iron treatment history
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Participants
  ≥1 course of intravenous iron | 24
  not received previous IV | 22
  unkown | 13

16. Secondary Outcome: Reason for Initiating Feraccru®
Description: Reason(s) for initiation of Feraccru®
Time Frame: Baseline
Population: The initiation reasons are not exclusive per patient. Some subjects had multiple reasons for initiating Feraccru®.
Measure: Count of Units; unit: initiation reasons
Units Other Than Participants: initiation reasons
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Number analyzed (initiation reasons) | 92
initiation reasons
  Intolerance to ferrous sulphate | 22
  Intolerance to ferrous fumarate | 15
  Intolerance to ferrous gluconate | 18
  Intolerance to oral iron | 7
  Clinician decision | 6
  Not recorded | 11
  Other | 13

17. Secondary Outcome: Percentage of Patients Who Discontinue Feraccru®
Description: Percentage of patients who discontinue Feraccru® during the 12 weeks period
Time Frame: Baseline to week 12
Measure: Number; unit: percentage of participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
percentage of participants | 49

18. Secondary Outcome: Reason for Discontinuing Feraccru®
Description: Reasons for stopping will be collected as predefined common options and a free text field.
Time Frame: Baseline to week 12
Population: The categories are not mutually exclusive so a single subject could have multiple reasons listed.
Measure: Number; unit: percentage of participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
percentage of participants
  Abdominal pain | 12
  Clinician decision | 5
  Diarrhoea | 3
  Constipation | 3
  Treatment complete | 3
  Lack of efficacy | 2
  Nausea | 2
  Not known | 17
  Other | 5

19. Secondary Outcome: Adverse Events That Are Related to and Caused by Feraccru®
Description: Type, severity and time of adverse events that are related to and caused by Feraccru®, from initiation of Feraccru®
Time Frame: For the duration of study, average of 12 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Participants
  definitely related | 1
  probably related | 7
  possibly related | 9

20. Secondary Outcome: Reason for Discontinuing Each Prior Oral Ferrous Product
Description: Reason(s) for discontinuing each prior Oral Ferrous Product (OFP). Patients could have multiple reasons for discontinuation of previous OFP.
Time Frame: Baseline
Population: Each discontinuation reason is exclusive per patient. Some patients had multiple reason for discontinuation.
Measure: Number; unit: individual reasons
Units Other Than Participants: individual reasons
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Number analyzed (individual reasons) | 34
individual reasons
  Diarrhoea | 4
  Nausea | 3
  Not known | 6
  Lack of efficacy | 8
  Treatment completion | 4
  Constipation | 1
  Flatulence | 1
  Abdominal pain | 3
  Unable to tolerate | 3
  Dramatically worsened GI symptoms | 1

21. Other Pre Specified Outcome: Sex of Patient at Baseline
Description: Sex of patient at Baseline - Male or Female
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Participants
  Male | 21
  Female | 38

22. Other Pre Specified Outcome: Type of IBD at Baseline (Crohn's Disease or Ulcerative Colitis)
Description: Type of Inflammatory Bowel Disease at baseline (Crohn's Disease or Ulcerative Colitis)
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 59
Participants
  Chron's Disease | 28
  Ulcerative Colitis (UC) | 28
  Unspecified IBD | 3

23. Other Pre Specified Outcome: Platelets Count at Baseline
Description: Mean platelets count at baseline
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 56
cells*10^9/L | 370.7 (131.4)

24. Other Pre Specified Outcome: Vitamin B12 Value at Baseline
Description: Vitamin B12 mean value at baseline
Time Frame: Baseline
Population: Subjects with available B12 measurement at Baseline.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 23
pmol/L | 354.6 (266.7)

25. Other Pre Specified Outcome: Mean Corpuscular Volume at Baseline
Description: Mean value of C-reactive protein (CRP) at Baseline
Time Frame: Baseline
Population: Subjects with available CRP value at Baseline
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 41
mg/L | 11.9 (18.0)

26. Other Pre Specified Outcome: Mean Corpuscular Hb at Baseline
Description: Mean corpuscular haemoglobin (MCH) at Baseline
Time Frame: Baseline
Population: 53 patients had MCH measured at Baseline.
Measure: Mean (Standard Deviation); unit: pg/cell
Arm/Group | Number of Eligible Subjects
Number analyzed (Participants) | 53
pg/cell | 27.0 (8.3)

ADVERSE EVENTS:
Time Frame: Baseline to approximately 12 weeks (permitting 10-16 weeks)
Arm/Group | Number of Eligible Subjects
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 1/59
Other Adverse Events (participants affected / at risk) | 9/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Eligible Subjects (N=59)
Right side buccal space abscess; (Infections and infestations) | 1 (1) — Right side buccal space abscess; admitted to hospital and treated.
Lower abdominal abscess (Gastrointestinal disorders) | 1 (1) — Lower abdominal abscess (secondary to CD)
Patient commenced with HB of 7.2 (Blood and lymphatic system disorders) | 1 (1) — Patient commenced on Feraccru® with HB of 7.2
gastritis and abdominal pain (Gastrointestinal disorders) | 1 (1) — Patient admitted overnight with gastritis and abdominal pain
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Number of Eligible Subjects (N=59)
Diarrhoea (Gastrointestinal disorders) | 6 (6) — Diarrhoea
Constipation (Gastrointestinal disorders) | 3 (3) — Constipation

LIMITATIONS AND CAVEATS:
Multiple patients lacked Hb (and other clinical parameters) at the 3-5- and 10-16-week time points, limiting the analysis that could be performed; due to this, overestimation or underestimation of the true normalisation rates may have been observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT03247816/Prot_SAP_000.pdf